CLINICAL TRIAL: NCT05415839
Title: Efficacy of Fractional CO2 Laser Versus Pulsed Dye Laser in the Treatment of Fingernail Psoriasis, a Randomized Controlled Trial.
Brief Title: Fractional CO2 Laser Versus Pulsed Dye Laser in Nail Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laser in nail psoriasis
Record Dates: First submitted 2022-01-07; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: the Efficacy of Fractional Co2 Laser in Nail Psoriais
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed dye laser (Active Comparator): Laser device
  Interventions: Device: Laser
- Fractional CO2 (Active Comparator): Laser Device
  Interventions: Device: Laser

INTERVENTIONS:
Device: Laser — Laser

SUMMARY:
The aim of this work is to assess the efficacy and safety of fractional CO2 laser therapy in comparison to pulsed dye laser (PDL) in the treatment of nail psoriasis.

DETAILED DESCRIPTION:
Study Design:

Randomized Clinical Trial

* Inclusion criteria:
* All patients with bilateral nail psoriasis.
* Age: Above 18
* Sex: both sexes
* Exclusion criteria:
* Cases who received treatment (systemic or topical) in the last 3 months before inclusion.
* Patients with proven onychomycosis by the microscopic mount of nail scraping
* Patients with excessive manual work
* Methodology in detail:
* All patients will be given written informed consent to participate in this study, children's parents are to sign their consent.
* Intra-patient randomization of 30 patients will be done so that the nails of each hand will be randomly included in one of two groups:

  1. Group A: The patient will receive 3 sessions of 1 month in-between of fractional CO2 laser with the following parameters: Two passes of 15 J, stacking 2, dwell time 500 Us, spacing 300 Um
  2. Group B: The patient will receive 3 sessions of pulsed dye laser of 1 month in-between with the following parameters: Two passes of 7 mm handpiece, 7.5 J, 0.5 msec pulse duration.
* Assessment will be carried as follows:

  * Full medical history of the disease and associated DM, HTN, or other systemic diseases.
  * Nail scrapping will be don by 30% KOH solution to exclude onychomycosis.
  * Clinical assessment by nail psoriasis index (NAPSI) (11) before treatment, 1 month and 3 months after the last session.
  * Photography before treatment, before each session of laser together with 1 month after the last session, and after 3 months of follow-up, photos will be examined by 2 blinded investigators.
  * Onychoscopic assessment will be done before treatment and after 1 month of the last session together with after 3 months follow up.
  * Capillorscopy of the proximal nail fold will be done before treatment and after 1 month of the last session together with after 3 months follow up.
  * Nail psoriasis quality of life scale (NPQ10) (12). will be done at the first visit, 1 month after the last session together with after 3 months follow up.
  * Visual analog scale (VAS) will be used to assess the pain of laser sessions.
  * Patient satisfaction will be reported at the end of the study by patient satisfaction score (excellent, very good, good, bad, very bad).
* Primary outcomes (Most important measurable outcomes)

  1. Assessment of the efficacy of fractional CO2 laser in the treatment of nail psoriasis clinically by photography and NAPSI score
  2. Comparing the safety and efficacy of fractional CO2 laser to the main type of laser used in nail psoriasis; PDL
* Secondary outcome parameters (other outcomes to be assessed)

  1. Onychoscopic assessment of the efficacy of fractional laser in treating nail psoriasis
  2. Determining the effect of fractional CO2 laser on both nail matrix and nail bed signs
  3. Capillorscopic assessment of both PDL and fractional CO2 laser on nail psoriasis

ELIGIBILITY:
Inclusion Criteria:

* - All patients with bilateral nail psoriasis.
* Age: Above 18
* Sex: both sexes

Exclusion Criteria:

* - Cases who received treatment (systemic or topical) in the last 3 months before inclusion.
* Patients with proven onychomycosis by the microscopic mount of nail scraping
* Patients with excessive manual work

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-25 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Nail psoriasis index (NAPSI) | change rom baseline at 3 months

SECONDARY OUTCOMES:
diameter of vessels by dermoscopy | change from baseline at 3 months